CLINICAL TRIAL: NCT01797198
Title: An Open Label, Drug-drug Interaction Study to Assess the Effect of Multiple Doses of Gemfibrozil on the Single Dose Pharmacokinetics of ASP3652 and to Assess the Effect of Multiple Doses of ASP3652 on the Single Dose Pharmacokinetics of Repaglinide
Brief Title: A Study to Assess the Effect of Multiple Doses of Gemfribozil on a Single Dose of ASP3652, and to Assess the Effects of Multiple Doses of ASP3652 on a Single Dose of Repaglinide in the Body of Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3652-CL-0006; 2011-002874-21 (EudraCT Number)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Drug-Drug Interaction (DDI); Healthy Subjects
Keywords: Phase I; ASP3652; Gemfibrozil; Repaglinide; Pharmacokinetics
MeSH Terms: interventions — ASP3652; Gemfibrozil; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gemfibrozil + ASP3652 (Experimental): Multiple doses of gemfibrozil and single dose of ASP3652
  Interventions: Drug: ASP3652; Drug: Gemfibrozil
- ASP3652 + repaglinide (Experimental): Multiple doses of ASP3652 and the single dose of repaglinide
  Interventions: Drug: ASP3652; Drug: Repaglinide

INTERVENTIONS:
Drug: ASP3652 — Oral
Drug: Gemfibrozil — Oral
  Arms: gemfibrozil + ASP3652
Drug: Repaglinide — Oral
  Arms: ASP3652 + repaglinide

SUMMARY:
ASP3652 is being investigated as a novel treatment for chronic pelvic pain. This is a two-part study to investigate the drug-drug potential of ASP3652.

Part I of the study evaluates the effect of gemfibrozil twice daily on the single dose of ASP3652.

Part 2 evaluates the effect of multiple doses of ASP3652 twice daily on the single dose of repaglinide.

Subjects participating in one part of the study may not participate in the other part.

DETAILED DESCRIPTION:
Part 1:

On Day 1, a single dose of ASP3652 is administered. After a wash-out period of 3 days, bid (twice daily) dosing of gemfibrozil starts on Day 4 and continues for 7 days until Day 10. On Day 8 (the 5th day of gemfibrozil administration), a single dose of ASP3652 is administered one hour after the morning dose of gemfibrozil.

Part 2:

On Day 1, a single dose of repaglinide is administered. After a wash-out period of 3 days, bid dosing of ASP3652 starts on Day 4 and continues for 7 days until Day 10. On Day 8 (the 5th day of ASP3652 administration), a single dose of repaglinide is administered one hour after the morning dose of ASP3652.

ELIGIBILITY:
Inclusion Criteria:

* Subject is white and of Caucasian origin.
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Male subjects must agree to practice an effective contraceptive method with female sexual partners to prevent pregnancy.

Exclusion Criteria:

* Known or suspected hypersensitivity to ASP3652, repaglinide and/or gemfibrozil, or any components of the formulation used.
* Any of the liver function tests (ALT, AST, γ-GT, TBL and ALP) above the upper limit of normal. In such case the sample may be repeated once.
* Regular use of any inducer of metabolism (e.g. barbiturates, Rifampicin) in the 3 months prior to admission to the Clinical Unit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of gemfibrozil on the Pharmacokinetics (PK) of a single dose of ASP3652 (plasma) and metabolites H1/H2/H3 | Days 1 - 11
  Part 1: Maximum concentration (Cmax), AUClast and AUCinf
Effect of multiple doses of ASP3652 on the PK of a single dose of repaglinide and metabolite M4 (plasma) | Days 1 - 10
  Part 2: Cmax, AUClast, AUCinf, and the ratio AUC(M4) / AUC(repaglinide)
Assess the safety of single and multiple doses of ASP3652 alone and in combination with gemfibrozil or repaglinide | Screening - End of Study Visit (7-14 days after (early) discharge)
  Both Parts: Vital signs, physical examination, adverse events, electrocardiogram, clinical laboratory assessments, body temperature, Bond and Lader Visual Analogue Scale (VAS) questionnaire, Physician's Withdrawal Checklist (PWC)

SECONDARY OUTCOMES:
Effect of multiple doses of gemfibrozil on the PK of a single dose of ASP3652 (plasma), metabolites H1/H2/H3 and Parent gemfibrozil and gemfibrozil-1-O-ß-glucuronide (plasma) | Days 1-11
  Part 1: tmax, tlag, t1/2, Vz/F, CL/F, Cmax, morning and evening Ctrough, tmax, AUCtau and CL/F
Effect of multiple doses of ASP3652 on the PK of a single dose of repaglinide | Days 1-10
  Part 2: tmax, tlag, t1/2, Vz/F, CL/F, Cmax, morning and evening Ctrough, tmax, AUCtau and CL/F
Effect of ASP3652 on the Pharmacodynamics (PD) of repaglinide by comparing the effect of repaglinide on blood glucose levels in the presence and absence of ASP3652 | Days 1-10
  Part 2: Baseline blood glucose concentration, minimum blood glucose concentration, and mean blood glucose concentration from 0 to 9h after dosing of repaglinide

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- PAREXEL Early Phase Clinical Unit, Harrow, United Kingdom